CLINICAL TRIAL: NCT06720506
Title: Comparsion Between Intrathecal Fentanyl and Intravenous Nalbuphine As a Postoperative Analgesia in Lower Limb Surgeries
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Khaled Helmy Abdelbasser, resident doctor at Anathesia and icu department Faculty of Medicine, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: fentanyl Vs nalbuphine LL surg
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Lower Limb Surgery
Keywords: fentanyl; nalbuphine
MeSH Terms: interventions — Fentanyl; Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group F (Experimental): patients will received intrathecal with dose 10-20ug
  Interventions: Drug: fentanyl
- group N (Experimental): Nalbuphine will given IV as shot in. Dose 1mg /kg
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Drug: fentanyl — Fentanyl will be given intrathecal with dose 10-20ug
  Arms: group F
Drug: Nalbuphine — Nalbuphine will given IV as shot in Dose 1mg /kg
  Arms: group N

SUMMARY:
Postoperative pain management has been a major challenge and there has been great interest about it ., there have been persistent efforts to bring out the best possible analgesic technique with the least side effects. The popularity of lower limb surgeries owing to its higher incidence, orthopedic and vascular surgerise. Inadequate postoperative pain relief is associated with undesirable side effects resulting in chronic persistent pain, delayed recovery Concern about opioid has powerful effect in relief post operative pain.

the aim of this study is to Compare between fentanyl intrathecal and nalbuphine IV as a postoperative analgesia in lower limb surgeries

DETAILED DESCRIPTION:
Fentanyl, a potent lipid-soluble opioid which was first synthesized more than 40years ago, is still the most popular opioid used as post operative analgesia t. Fentanyl given intrathecally use in many acute and chronic pain conditions. inspite of its side effects fentanyl remains the mainstay of anesthesiologists in post operative period analgesia.

Anesthetic methods of Lower limb surgery such as orthopedic and vascular surgeries, for example in the use of local infiltration, spinal anesthesia, caudal anesthesia, or general anesthesia Among them, spinal anesthesia is commonly used for lower limb surgery which does not need a sophisticated machine and which has been performed for years before anesthetic equipment such as mechanical ventilators and monitoring devices was produced. The development of new local anesthetic agents, the use of opioids, and an interest in acute and chronic pain management have universalized spinal anesthesia. Immediate pain is very severe in lowerlimb surgery and difficul to control. Moreover, due to the short hospitalization period, there is a limit in the application of patient-controlled analgesia that permits patients to treat pain by directly activating doses of opoids .

Nalbuphine...

Nalbuphine is an agonist-antagonist opioid and provides prolonged duration of analgesia with

fewer side effects of fentanyl such as pruritus, nausea, and vomiting.

Nalbuphine has a powerful effect in decreasing postoperative pain nNalbuphine IS asynthetic agonistant agonist opioid, demonstrated to attenuate mu-opioid receptor-related adverse events such as pruritis, nausea/emesis, constipation respiratory depression, undesirable sedation, and the development of toler ance and dependence. With several clinical reports, nalbuphine has been recognized as a safe and highly efficacious opioid analgesic that possesses remarkably low narcotic abuse liability. As a result, nalbuphine provides an alternative choice to replace strong opioids for the clinical practice of post- operative pain managemen

ELIGIBILITY:
Inclusion Criteria:

* male and female pt between 18 and 600 year
* pt with lower limb surgeries with no. Indication for general anathesia
* patient with no contraindication for spinal anatthesia

Exclusion Criteria:

* pt who refuses
* pt with hypersensivity to any drug
* pt addicts opiods
* chronic use of opiod
* Inability to comprehend postoperatively the pain assessment scale/neuropsychiatric disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
first request of rescue analgesia | 24 hours
  Duration of analgesia until first analgesic request

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Culebras X, Gaggero G, Zatloukal J, Kern C, Marti RA. Advantages of intrathecal nalbuphine, compared with intrathecal morphine, after cesarean delivery: an evaluation of postoperative analgesia and adverse effects. Anesth Analg. 2000 Sep;91(3):601-5. doi: 10.1097/00000539-200009000-00019. PMID 10960384
- [Background] Pick CG, Paul D, Pasternak GW. Nalbuphine, a mixed kappa 1 and kappa 3 analgesic in mice. J Pharmacol Exp Ther. 1992 Sep;262(3):1044-50. PMID 1326621